CLINICAL TRIAL: NCT04584385
Title: Advanced EEG Technology in Childhood Epilepsy: A Multimodal Wearable Approach for Long-term Seizure Detection and Sleep Monitoring.
Brief Title: Advanced EEG Technology in Childhood Epilepsy
Acronym: PnP
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Byteflies (Industry)
Responsible Party: Sponsor
Other Study IDs: s64658
Record Dates: First submitted 2020-09-23; First posted 2020-10-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy in Children; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Childhood epilepsy: Children with refractory tonic, myoclonic or atonic seizures
  Interventions: Diagnostic Test: EEG

INTERVENTIONS:
Diagnostic Test: EEG — EEG monitoring

SUMMARY:
A lot of effort has already been put into the development of smaller, wearable and more user-friendly devices to monitor seizures in patients with epilepsy.

The investigators hypothesize that a wearable EEG ( in combination with additional non-EEG biosignals (motion, ECG, EMG, respiration, temperature,...) derived from Byteflies Sensor Dot and new medical patches (Plug 'n Patch system), will be able to objectively detect epileptic seizures and monitor sleep in the hospital and home environment for specific types of childhood epilepsy.

The accuracy of seizure detection and sleep monitoring by the wearable miniature EEG device in combination with other (autonomic) biosignals (full PnP system) will be compared with the golden standard video-EEG and seizure and sleep diaries filled-out by the participants.

DETAILED DESCRIPTION:
The objective of the study will be the following:

1. Multimodal seizure detection Evaluation of data quality and seizure annotation accuracy. Comparison of data derived from the multimodal wearable device (Sensor dot in combination with Plug and Patch system) versus video EEG and seizure diary in childhood epilepsy syndromes with

   * Tonic seizures
   * Atonic seizures
   * Myoclonic seizures During wakefulness and during sleep
2. Sleep monitoring Assessment of sleep data quality, latency, sleep fragmentation and time spent in different sleep stages in different childhood epilepsy syndromes. Investigation of the influence of occuring seizures on sleep architecture.

Comparison of data wearable device (Byteflies Sensor Dot in combination with Plug and Patch system) versus video-EEG and sleep diary in childhood epilepsy syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Childhood epilepsy with tonic, atonic or myoclonic seizures
* Parental informed consent and assent of the child if applicable
* Parent or caregiver can keep a seizure and sleep diary reliably.

Exclusion criteria

* Inability to provide written informed consent by parent or caregiver.
* Known allergy to electrodes or medical adhesives used as part of the study protocol.
* Having an implanted device, such as (but not limited to) a pacemaker, ICD, VNS because Sensor Dot contains magnets that could interfere with the operation of these devices.
* Any other condition or finding that would compromise the safety of the participant or the quality of the study data, or otherwise interfere with achieving the study objectives, as determined by the investigator or research coordinator.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between 4 and 18 years old with epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of seizure detection in-hospital | 24 hours
  Accuracy (F1 score, precision and recall) of wearable multimodal device for seizure detection. Comparison of data with golden standard video EEG.
Accuracy of sleep monitoring in-hospital | 24 hours
  Assessment of sleep parameters with wearable multimodal device. Comparison of data with golden standard video EEG. Sleep scoring will be done according to American Academy of Sleep Medicine.

SECONDARY OUTCOMES:
Accuracy of seizure detection at home | 1-21 days
  Accuracy of wearable multimodal device for seizure detection versus seizure diary filled out by the participant or caregiver.
Accuracy of sleep monitoring at home | 1-21 days
  Accuracy of sleep monitoring of the wearable multimodal device versus sleep checklist (Sleep Behavior Questionnaire (SQ-SP A.P.H.M. Maas, W. Braam, R. Didden, M. Smits, & L.M.G. Curfs 2005 )

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Proost R, Heremans E, Lagae L, Van Paesschen W, De Vos M, Jansen K. Automated sleep staging on reduced channels in children with epilepsy. Front Neurol. 2024 May 10;15:1390465. doi: 10.3389/fneur.2024.1390465. eCollection 2024. PMID 38798709